CLINICAL TRIAL: NCT04787692
Title: Impact of Daily, Digital and Behavioral Tele-health Tapering Program for Perioperative Surgical Patients Exposed to Opioids and Benzodiazepines.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Evan Pivalizza, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-0549
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Elective Spine Surgery Receiving Pre and/or Postoperative Pain Control With Opioids
Keywords: Opioid taper; post-surgery; behavioral tele-health
MeSH Terms: interventions — Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid and Benzodiazepine Naive-patients (Experimental): Opioid and Benzodiazepine Naive-patients, defined as no medications 30 days prior to surgery
  Interventions: Behavioral: Opioid and Benzodiazepine Naive-patients
- Opioid and Benzodiazepine Tolerant-patients (Experimental): Opioid and Benzodiazepine Tolerant-patients, defined as use of medications on most days for 1 or more months (>30 days) prior to surgery
  Interventions: Behavioral: Opioid and Benzodiazepine Tolerant-patients

INTERVENTIONS:
Behavioral: Opioid and Benzodiazepine Naive-patients — Duration of treatment : 1 month Lucid Lane is a service that will be used by patients scheduled for elective orthopedic or neurosurgical spine surgery that will incorporate continuous MEASUREMENT & MONITORING, PERSONALIZED TREATMENT PLANNING and REAL-TIME INTERVENTIONS (MPI) as the patient is tapering off of opioids and/or benzodiazepines. Patients will participate in the Lucid Lane program.Daily support will include 1 or more from the following: Therapist chat, and/or audio psychotherapy sessions, and/or group therapy sessions, Cognitive behavioral therapy(CBT), Mindfulness, and/or peer support. Patients will submit a weekly survey and the therapist will submit weekly reports to the physician.
  Arms: Opioid and Benzodiazepine Naive-patients
Behavioral: Opioid and Benzodiazepine Tolerant-patients — Duration of treatment : 6 months Lucid Lane is a service that will be used by patients scheduled for elective orthopedic or neurosurgical spine surgery that will incorporate continuous MEASUREMENT & MONITORING, PERSONALIZED TREATMENT PLANNING and REAL-TIME INTERVENTIONS (MPI) as the patient is tapering off of opioids and/or benzodiazepines. Patients will participate in the Lucid Lane program.Daily support will include 1 or more from the following: Therapist chat, and/or audio psychotherapy sessions, and/or group therapy sessions, CBT, Mindfulness, and/or peer support. Patients will submit a weekly survey and the therapist will submit weekly reports to the physician.
  Arms: Opioid and Benzodiazepine Tolerant-patients

SUMMARY:
The purpose of this study is to examine the safety, acceptability, and feasibility of a controlled taper off of opioids and/or benzodiazepines, with the use of behavioral health tele-health based therapy services, in the perioperative patient.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative benzodiazepines opioid dependence (daily use of opioids or benzodiazepines preoperatively) (Naive: No Meds 30 Days Prior to surgery,Opioid tolerant/dependant: Use of Meds on Most Days For 1 or more months prior to surgery)
* Subject willing to use Lucid Lane program to provide behavioral health support perioperative period up to 6 months post-op for tolerant opioid/benzo users
* Subject is willing to discuss Lucid Lane progress with the University of Texas Health Science Center(UTHealth) perioperative team and prescribing clinicians
* Subject is willing to sign a Lucid Lane Client Agreement
* Willing to sign an informed consent

Exclusion Criteria:

* Serious mental illnesses including schizophrenia-spectrum disorders, severe bipolar disorder, and severe major depression.
* Active suicidal ideations
* Patients on methadone or buprenorphine for treatment of opioid use disorder (i.e. for treatment of addiction, and not for treatment of pain)
* Patient unwilling to use or not possessing access to a device that allows for video visits (e.g. a smartphone, tablet, or computer)
* Patients who are on palliative care
* Insufficient ability to use English to participate in the consent process, the intervention or study assessments.
* Insufficient ability to provide informed consent to participate
* If the patient misses more than 2 lucid lane sessions per week, the staff will be immediately notified by Lucid Lane.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of patients that engage and participate in the process | 30 days post intervention
  Engagement and participation are defined as patient's commitment for 1 hour a week as scheduled.
Number of patients that engage and participate in the process | 90 days post intervention
  Engagement and participation are defined as patient's commitment for 1 hour a week as scheduled.
Number of patients that engage and participate in the process | 180 days post intervention
  Engagement and participation are defined as patient's commitment for 1 hour a week as scheduled.

SECONDARY OUTCOMES:
Percentage of patients in the naive group that successfully taper off of the benzodiazepine or opioid | 30 days post intervention
Percentage of patients in the naive group that successfully taper off of the benzodiazepine or opioid | 90 days post intervention
Percentage of patients in the tolerant group that successfully taper off of the benzodiazepine or opioid | 180 days post intervention
Emotional well-being as measured by the Generalized Anxiety Disorder 7-item (GAD-7) scale | 30 days post intervention
  The Generalized Anxiety Disorder 7-item (GAD-7) scale has 7 questions each ranging in score from 0-3, with a higher score indicating a worse outcome.
Emotional well-being as measured by the The Patient Health Questionnaire 9 (PHQ-9) | 30 days post intervention
  The Patient Health Questionnaire 9 (PHQ-9) consists of 10 questions with a total score ranging form 1 to 27, with a higher score indicating greater depression.
Symptoms as measured by the Edmonton Symptom Assessment System (ESAS) | 30 days post intervention
  The Edmonton Symptom Assessment System consists of 10 questions, each question ranging from 0-10, with a higher score indicating a worse outcome. The ESAS rates the intensity of common symptoms, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath.
Emotional well-being as measured by the Generalized Anxiety Disorder 7-item (GAD-7) scale | 90 days post intervention
  The Generalized Anxiety Disorder 7-item (GAD-7) scale has 7 questions each ranging in score from 0-3, with a higher score indicating a worse outcome.
Emotional well-being as measured by the Patient Health Questionnaire 9 (PHQ-9) | 90 days post intervention
  The Patient Health Questionnaire 9 (PHQ-9) consists of 10 questions with a total score ranging form 1 to 27, with a higher score indicating greater depression.
Well-Being as measured by the Edmonton Symptom Assessment System (ESAS) | 90 days post intervention
  The Edmonton Symptom Assessment System consists of 10 questions, each question ranging from 0-10, with a higher score indicating a worse outcome. The ESAS rates the intensity of common symptoms, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath.
Emotional well-being as measured by the Generalized Anxiety Disorder 7-item (GAD-7) scale | 180 days post intervention
  The Generalized Anxiety Disorder 7-item (GAD-7) scale has 7 questions each ranging in score from 0-3, with a higher score indicating a worse outcome.
Emotional well-being as measured by the Patient Health Questionnaire 9 (PHQ-9) | 180 days post intervention
  The Patient Health Questionnaire 9 (PHQ-9) consists of 10 questions with a total score ranging form 1 to 27, with a higher score indicating greater depression.
Well-Being as measured by the Edmonton Symptom Assessment System (ESAS) | 180 days post intervention
  The Edmonton Symptom Assessment System consists of 10 questions, each question ranging from 0-10, with a higher score indicating a worse outcome. The ESAS rates the intensity of common symptoms, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath.
Quality of life as measured by the Quality of life Score | 30 days post intervention
  The range of scores is between 15 to 105, with a higher score or number being indicative of a higher quality of life.
Quality of life as measured by the Quality of life Score | 90 days post intervention
  The range of scores is between 15 to 105, with a higher score or number being indicative of a higher quality of life.
Quality of life as measured by the Quality of life Score | 180 days post intervention
  The range of scores is between 15 to 105, with a higher score or number being indicative of a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Evan G Pivalizza, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hussain M, Norgeot B, Zaafran A, Stark J, Caridi J, Fenoy A, Pivalizza E. Virtual transitional pain service delivered via telehealth is effective in preventing new and persistent opioid use amongst post-surgical spine patients. medRxiv [Preprint]. 2023 Aug 20:2023.08.18.23294272. doi: 10.1101/2023.08.18.23294272. PMID 37645940